CLINICAL TRIAL: NCT03430947
Title: An Open-label Phase II Multicenter Study of Vemurafenib (Zelboraf®) Plus Cobimetinib (Cotellic®) After Radiosurgery in Patients With Active BRAF-V600-mutant Melanoma Brain Metastases
Brief Title: Vemurafenib Plus Cobimetinib After Radiosurgery in Patients With BRAF-mutant Melanoma Brain Metastases
Acronym: RadioCoBRIM
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to insufficient recruitment, the clinical trial was terminated prematurely
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TUD-CoBRIM-67; 2017-000768-13 (EudraCT Number)
Record Dates: First submitted 2018-01-10; First posted 2018-02-13 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Malignant Melanoma Stage IV; BRAF V600 Mutation; Brain Metastases
Keywords: Stereotactic radiosurgery; BRAF inhibitor; MEK inhibitor; Vemurafenib; Cobimetinib
MeSH Terms: conditions — Melanoma; Brain Neoplasms | interventions — Vemurafenib; cobimetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): all patients will be treated with Vemurafenib + Cobimetinib
  Interventions: Drug: Vemurafenib; Drug: Cobimetinib

INTERVENTIONS:
Drug: Vemurafenib — Vemurafenib (960 mg twice a day) will be taken on days 1 - 28 of each 28-day treatment cycle.
Drug: Cobimetinib — Cobimetinib (60 mg once a day) will be taken on days 1 - 21 of each 28-day treatment cycle.

SUMMARY:
This is a phase II, open label, non-randomised study of vemurafenib and cobimetinib after radiosurgery in adult patients with BRAFV600-mutant melanoma brain metastases. All patients will receive vemurafenib 960 mg twice a day on days 1 - 28 combined with cobimetinib 60 mg once a day on days 1 - 21 of each 28-day treatment cycle until disease progression, drug toxicity or death.

The primary objective of this study is to determine the best overall response rate (BORR) in the brain. The extracranial BORR, intra- and extracranial duration of response, progression-free survival and overall survival, adverse events, quality of life and radiomics features predicting long-term local control of brain metastases and treatment-related toxicity will also be examined.

ELIGIBILITY:
Inclusion criteria

* Signed informed consent
* Female and male patients ≥ 18 years of age
* Histologically confirmed metastatic melanoma (stage IV, per AJCC staging), carrying BRAF V600-mutation
* Performed SRS 14 ±7 days before baseline using a harmonized protocol in patients with at least one measurable intracranial target lesion for which the following criteria are met:

  * Previously untreated (Lesions in previously irradiated area should not be selected)
  * Largest diameter of ≥ 0.5 but ≤ 4 cm as determined by contrast-enhanced MRI and
  * ≤ 10 brain metastases
* ECOG performance status 0 - 2
* Life expectancy ≥ 12 weeks
* Adequate bone marrow function as indicated by the following:

  * ANC ≥ 1500/µL,
  * Platelets ≥ 100,000/µL and
  * Hemoglobin ≥ 9 g/dL
* Adequate renal function, as indicated by creatinine ≤ 1.5 x ULN
* Adequate liver function, as indicated by bilirubin < 1.5 x ULN and AST and ALT < 3 x ULN (documented liver metastases: AST and ALT < 5 x ULN)
* Adequate coagulation within 28 days prior to baseline visit

  * Patients without therapeutic anticoagulation: INR or aPTT ≤ 1.5 x ULN
  * Patients receiving therapeutic anticoagulation: stable anticoagulation regimen and stable INR
* Able to swallow pills

Exclusion criteria

* Symptomatic brain metastases requiring immediate local interventions such as neurosurgery or radiosurgery
* Leptomeningeal disease (also synchronous with brain metastases)
* Prior therapy with BRAF or MEK inhibitors within 12 weeks prior to baseline visit (prior therapies for metastatic melanoma including chemo-, cytokine-, immuno-, biological and vaccine-therapy will be al-lowed) A period of at least 6 weeks must be observed between the last dose of ipilimumab and the first administration of the study treatments. Prior treatment with anti-programmed cell death (PD)-1 or anti-PD ligand 1 (PD-L1) is allowed.
* Prior whole brain irradiation (Patients with prior local therapy of brain metas-tases are eligible)
* Patients receiving therapeutic steroids are not stable on corticoster-oids 2 weeks before SRS
* Active and uncontrolled infection
* Known HIV infection or active HBV or HCV infection

  * Active HBV infection (chronic and acute), defined as having a posi-tive hepatitis B surface antigen (HBsAg) test at screening (past or resolved HBV infection, defined as negative HBsAg test and a posi-tive total hepatitis B core antibody test at screening, are eligible)
  * Active HCV infection, defined as positive HCV antibody test and positive HCV RNA test at screening
* Intracranial radiation therapy within 14 days prior to SRS
* Extracranial radiation therapy within the last 14 days prior to baseline visit
* Treatment with strong CYP3A4/5 inhibitors (e.g. ketoconazole) and inducers (e.g. phenytoin, carbamazepine). (anticonvulsant levetiracetam is allowed; patient should be stable on levetiracetam for 2 weeks)
* Unresolved toxicity of National Cancer Institute Common Terminology Crite-ria for Adverse Events, version 4.0 (NCI v4.0) [NCI, 2009] Grade 2 or higher from previous anti-cancer therapy, except alopecia.
* Conditions that will interfere significantly with the absorption of drugs (e.g. Colitis ulcerosa)
* Inability to undergo MRI secondary to:

  * Metal,
  * Claustrophobia, or
  * Gadolinium contrast allergy
* Previous malignancies active within the last 3 years, with the exception of locally curable cancers that have been treated to complete remis-sion or untreated stage I chronic lymphoid leukemia.
* Unwillingness or inability to comply with study and follow-up procedures
* Known hypersensitivity to any of the excipients of cobimetinib and vemuraf-enib
* The following foods/supplements are prohibited at least 7 days prior to initia-tion of and during study treatment:

  * St. John's wort or hyperforin (potent cytochrome P450 CYP3A4 enzyme inducer)
  * Grapefruit juice (potent cytochrome P450 CYP3A4 enzyme inhibitor)
* Patient is included in another interventional trial
* Use of any investigational or non-registered product within 4 weeks prior to baseline visit
* Woman of childbearing age with the exception they meet at least one of the following criteria:

  * Post-menopausal,
  * Sterilization,
  * Consistently & correct application of contraceptives (Pearl Index < 1%),
  * sexual abstinence, or
  * vasectomy of the partner
* Pregnant or lactating women
* History, risk factor or retinal pathology that increases the risk of retinal vein occlusion (RVO) or central serous retinopathy (CSR): evidence of retinal pathology that is considered a risk factor for RVO or CSR, or a history of retinal detachment, central serous chorioretinopathy or reti-nal vein thrombosis. The risk factors for RVO are listed below:

  * Uncontrolled glaucoma with intraocular pressures > 21 mm Hg,
  * Serum cholesterol ≥ Grade 2 (≥ 7.75 mmol/L),
  * Hypertriglyceridemia ≥ Grade 2 (≥ 3.42 mmol/L), Hyperglycemia (fasting) ≥ Grade 2 (≥ 8.9 mmol/L).
* History of clinically significant cardiac dysfunction including:

  * Myocardial infarction,
  * Severe/unstable angina pectoris,
  * Symptomatic congestive heart failure (NYHA stage ≥ 2),
  * cerebrovascular accident or transient ischemic attack within the previous 6 months,
  * History of congenital long QT syndrome or mean QTcF > 450 msec or uncorrectable electrolyte abnormalities,
  * Hypertension > Grade 2 not controlled by medications
  * Left ventricular ejection fraction (LVEF) < 50%, or
  * Uncontrolled arrhythmias

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
Best overall response rate in the brain | 2 years
  rate of patients with complete response or partial response (intracranial)

SECONDARY OUTCOMES:
Extracranial best overall response rate | 2 years
  rate of patients with complete response or partial response (extracranial)
Best overall response rate calculated for the whole body tumor sites | 2 years
  rate of patients with complete response or partial response
Intracranial duration of response | 2 years
  time from best overall response in the brain to first documentation of intracranial progression
Extracranial duration of response | 2 years
  time from best extracranial overall response to first documentation of extracranial progression
Progression-free survival | 2 years
  time from first dose of study treatment until progression
Overall survival | 2 years
  time from first dose of study treatment until death due to any cause
Incidence of adverse events | 2 years
  Adverse events by type, frequency and severity using National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 4.03; number of patients who withdraw from the study due to intolerable adverse events.
Radiomics for long-term control of brain metastases | every 6 weeks up to 2 years
  Radiomics features predictive of long-term local control of brain metastases using Magnetic Resonance Imaging
Radiomics for intracranial Treatment-related toxicity | every 6 weeks up to 2 years
  Radiomics features predicting treatment-related toxicity (e.g. radionecrosis, hemorrhage, edema) using Magnetic Resonance Imaging

CONTACTS AND LOCATIONS:
Overall Officials: Friedegund Meier, MD, Principal Investigator — Technische Universität Dresden
Locations (3):
- Germany (3):
  - Technische Universität Dresden, Dresden
  - Ruprecht-Karls-University of Heidelberg, Faculty of Medicine, Heidelberg
  - Eberhard Karls University of Tübingen, University Medical Center, Tübingen

IPD SHARING:
Plan to Share IPD: Yes
After publication of the primary objective, the data might be provided to interested scientists on request (e.g. for meta-analyses or other scientific research) in an anonymized way within 5 years (according to the General Data Protection Regulation), provided that the sponsor and the coordinating principal investigators have given their prior written consent.
Supporting Information: CSR
Time Frame: within 5 years